CLINICAL TRIAL: NCT05145660
Title: Optimization of Cervical Nodal Clinical Tumor Volume for Early and Medium Stage Nasopharyngeal Carcinoma: a Multicenter Non-inferior Randomized Controlled Phase III Clinical Trial
Brief Title: Optimization of Cervical Nodal CTV for Early and Medium Stage NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jun-Lin Yi, MD (Unknown)
Responsible Party: Sponsor-Investigator, Jun-Lin Yi, MD, Radiotherapy director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-2021C-257
Record Dates: First submitted 2021-11-12; First posted 2021-12-06 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Involved site irradiation (Experimental): High-risk CTV1 : GTVnx plus a 10-mm margin to encompass the microscopic extension of the gross tumor, the whole nasopharynx, the high-risk structures recommended for CTVp2 by the contouring consensus* (such as parapharyngeal space, skull base, pterygopalatine fossa and the inferior part of the nasal cavity and maxillary sinus), the VIIa, and the retrostyloid space above the bilateral transverse process of C1.
  Low-risk CTV2:
  N0/positive RPLN only: Bilateral cervical nodal region with the 3-cm caudal expansion below transverse process of C1, and at least covering the level II.
  N1-2 (positive cervical LNs): Ipilateral cervical nodal region with the 3-cm expansion below the positive LN (GTVnd), and at least covering the level II; contralateral cervical nodal region with the 3-cm caudal expansion below the transverse process of C1, and at least covering the level II.
  Suspicious LN: 1-cm expansion below the suspicious LN (GTVnd-suspicious)
  Interventions: Radiation: intensity-modulated radiotherapy (IMRT) with reduced-volume; Drug: Chemotherapy
- Elective region irradiation (Active Comparator): High-risk CTV1 : GTVnx plus a 10-mm margin to encompass the microscopic extension of the gross tumor, the whole nasopharynx, the high-risk structures recommended for CTVp2 by the contouring consensus* (such as parapharyngeal space, skull base, pterygopalatine fossa and the inferior part of the nasal cavity and maxillary sinus), the VIIa, and the retrostyloid space above the bilateral transverse process of C1.
  Low-risk CTV2:
  N0/positive RPLN only: Bilateral level III + Va N1-2 (positive cervical LNs): At least one subsequent level below CTV1
  Interventions: Radiation: intensity-modulated radiotherapy (IMRT) with reduced-volume; Drug: Chemotherapy

INTERVENTIONS:
Radiation: intensity-modulated radiotherapy (IMRT) with reduced-volume — PGTVnx: 69.9Gy/2.12Gy/33f GTVrpn: 69.9Gy/2.12Gy/33f GTVnd: 69.9Gy/2.12Gy/33f GTVnd-suspicious: 60.06Gy/1.82Gy/33f PTV1: 60.06Gy/1.82Gy/33f PTV2: 50.96Gy/1.82Gy/28f
  Other Names: intensity-modulated radiotherapy
Drug: Chemotherapy — Concurrent cisplatin (100 mg/m², d1-3, Q3w, maximum to three cycles); The application of induction chemotherapy and consolidation chemotherapy is dependent on the physician's discretion.

SUMMARY:
Current radiotherapy guidelines and consensus statements uniformly recommend elective region irradiation (ERI) as the standard strategy for nasopharyngeal carcinoma (NPC). However, given the scarcity of skip-metastasis, the improved assessment accuracy of nodal involvement, and the striking advancements in chemotherapy for NPC, a one-fits-all delineation scheme for clinical target volumes for the nodal region (CTVn) may not be appropriate anymore, and modifications of the CTVn delineation strategy may be warranted. Involved site irradiation (ISI) covering merely the initially involved nodal site and potential extranodal extension has been confirmed to be as effective as ERI with decreased radiation-related toxicities in some malignancies, but has not yet been investigated in NPC. This study aims to compare the regional control, survival outcomes, radiation-related toxicities, and quality of life (QoL) of ISI with conventional ERI in NPC patients with a limited nodal burden.

DETAILED DESCRIPTION:
ISRT-NPC is a prospective, multicenter, open-label, noninferiority, phase III randomized controlled trial. A total of 488 patients will be randomly assigned in a 1:1 ratio to receive ISI or ERI. Randomization will be stratified by institution and N stage. Generally, in the ISI group, the high-risk CTV1 (dose: 60 Gy) includes a 1-cm expansion of the positive LN as well as the VIIa and the retrostyloid space above the bilateral transverse process of the atlantoaxial spine (C1), regardless of N status. The low-risk CTV2 (Dose: 50 Gy) covers the cervical nodal region with a 3-cm caudal expansion below the transverse process of C1 for N0 disease and a 3-cm expansion below the positive LN for positive LNs (at least covering the level II).

ELIGIBILITY:
1. Age between 18 and 75 years;
2. Karnofsky performance status (KPS) score ≥ 70;
3. Pathologically confirmed World Health Organization (WHO) type II-III NPC;
4. TNM stage I-III (T1-3N0-2M0) according to the 8th American Joint Committee on Cancer / Union for International Cancer Control (AJCC/UICC) staging system with a maximum diameter (MAD) of cervical involved LNs ≤ 3 cm, namely LB-LN;
5. Available baseline nasopharynx and neck computed tomography (CT) or magnetic resonance imaging (MRI) (strongly advocated) data (including functional MRI sequences) and measurable tumor lesions;
6. All procedures for defining the tumor burden completed within 4 weeks of registration;
7. Survival expectancy of at least 6 months;
8. Normal marrow and organ function: hemoglobin ≥ 120 g/L, WBCs ≥ 4 × 109 /L, platelets ≥ 100 × 109 /L; liver and kidney function-related indicators within 1.25*the normal upper limit;
9. Patient willingness to comply with the protocol;
10. Patient willingness and ability to provide an informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Regional-recurrence-free survival | 3-year
  measured from the registration to the documented regional recurrence

SECONDARY OUTCOMES:
Overall survival | 3-year
  measured from registration to documented death from any cause or last follow-up
Distant metastasis-free survival | 3-year
  measured from registration to documented distant metastasis or death from any cause
Progression-free survival | 3-year
  measured from registration to documented locoregional recurrence or distant metastasis or death from any cause
Number of Participants with acute and late radiation-related toxicities | 8-year
  Acute radiation-related toxicities are assessed using the National Cancer Institute Common Toxicity Criteria version 4.0 scale. Acute radiation-related toxicities include dermatitis, mucositis, dry mouth, dysphagia, trismus, and subcutaneous soft tissue. Late radiation toxicities are assessed according to the Radiation Therapy Oncology Group (RTOG) and European Organisation for Research and Treatment of Cancer (EORTC) late radiation morbidity scoring scheme, including skin, neck tissue damage, hypothyroidism, dry mouth, dysphagia, trismus, and other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China

REFERENCES:
- [Derived] Liu Y, Han Y, Liu F, Hu D, Chen Z, Wang P, Li J, Qin J, Jin F, Li Y, Wang J, Yi J. Involved site radiation therapy in stage I-III nasopharyngeal carcinoma with limited lymph node burden (ISRT-NPC) or elective region irradiation: a study protocol for a multicenter non-inferiority randomized controlled phase III clinical trial. BMC Cancer. 2023 Aug 3;23(1):724. doi: 10.1186/s12885-023-11212-7. PMID 37537541